CLINICAL TRIAL: NCT04568460
Title: Standing Tall (Yima Nkqo): A Pilot Randomized Controlled Trial of a Community-Based Intervention to Improve Health Outcomes for Young Adults Newly Diagnosed With HIV in South Africa
Brief Title: Standing Tall (Yima Nkqo)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Desmond Tutu Health Foundation (Other); University of Connecticut (Other); Columbia University (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Ingrid Theresa Katz, M.D., Associate Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002671
Record Dates: First submitted 2020-08-12; First posted 2020-09-29 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Sessions (Experimental): Intervention group sessions will be delivered by lay health counselors. The sessions will reflect principles of co-learning, participatory design, and empowerment to promote engagement of young people in critical thinking and problem solving - including modeling, roleplaying, and interactive activities.
  Interventions: Other: Intervention Group Sessions
- Standard of Care (No Intervention): This is the standard of care arm. Participants newly diagnosed with HIV will get a referral to the local primary health care setting of their choice for further management, including ART.

INTERVENTIONS:
Other: Intervention Group Sessions — Participants will undergo a multi-session group intervention over the course of six months.
  Other Names: Yima Nkqo
  Arms: Intervention Group Sessions

SUMMARY:
The investigators propose the Standing Tall study, a prospective randomised study of strategy to optimize community-based ART initiation in South Africa. Investigators will work closely with community members to integrate community-based ART. One hundred participants will be enrolled and followed for a total of up to 6 months. Those in the intervention arm will be provided with the ST intervention which includes a behavioral component and access to ART. The intervention will be linked to a clinic through a "Nurse Initiated Management of ART."

DETAILED DESCRIPTION:
The premise for our study is based on three decades of HIV research that supports the need for multi-component, multisystem interventions to promote testing, and adherence to treatment and care for young people living with HIV. The proposed intervention, Standing Tall, is informed and guided by Social Action Theory - a conceptual framework reflecting a holistic understanding of health behavior and motivational factors that foster and maintain behavior change. Standing Tall, a pilot randomized controlled trial, is designed to address multi-factorial barriers using (1) a socio-behavioral group intervention; (2) social support; (3) provision of immediate ART and refills. The primary outcome is ART initiation at three months, and the secondary outcome is viral load suppression at six months. Other tertiary/exploratory outcomes include behavioral outcomes and process evaluation of the intervention itself, and the use of point-of-care diagnostics.

The administrative supplemental funding provides support for an additional objective of this study: to understand how best to use point-of-care (POC) testing in clinical practice in order to improve HIV care and treatment for South African young people. Understanding patient perspectives and perceived barriers is critical to developing feasible, acceptable, and effective protocols for implementing POC testing. The primary aim for achieving this objective is to assess patient perspectives regarding POC testing through in-depth, semi-structured interviews among study participants enrolled in Standing Tall's second aim.

ELIGIBILITY:
Inclusion Criteria:

* Complete an assessment of understanding
* Provide informed consent
* Are between ages 18-24
* Present to Tutu Tester vans in Cape Town OR East London DTHF clinics (Duncan Village Day Hospital, Empilweni Gompo Health Centre, Gompo C Clinic) and test HIV+
* Are ART-naïve
* Are English or isiXhosa speakers
* Reside in the Cape Town or East London metro area

Exclusion Criteria:

* Are pregnant (must be referred to antenatal clinic if living with HIV)
* Test positive for tuberculosis (must be referred to clinic for TB treatment prior to ART initiation)
* Are unable to understand the process of informed consent

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
ART Initiation | Three Months
  ART initiation will be assessed via a self-report measure of participants who will report whether they have or have not initiated ART.
ART Initiation | Three Months
  ART initiation will also be assessed via a point-of-care diagnostic detecting Tenofovir concentrations in participants.
ART Initiation | Six months
  ART initiation will be assessed via a self-report measure of participants who will report whether they have or have not initiated ART.
ART Initiation | Six months
  ART initiation will also be assessed via a point-of-care diagnostic detecting Tenofovir concentrations in participants.

SECONDARY OUTCOMES:
Viral Load Suppression | Six Months
  Viral suppression will be measured from plasma specimen collected at 6 months from enrollment. Persons missing plasma HIV RNA results for any reason (e.g. death) will be counted as not initiated. Additional records obtained through PHDC and NHLS will provide additional data (such as plasma HIV RNA concentration) that will be used for confirmation.
Household Food Security | Six Months
  We will assess household food security via a self-report questionnaire. Participants will report how many times in the last 30 days they experienced anxiety and uncertainty about household food access and insufficient quality and quantity on a scale from rarely to more than 10 times.
Mental Health | Six Months
  We will assess generalized anxiety disorder using the GAD-7 questionnaire and major depressive disorder using the Patient Health Questionnaire (PHQ-9). Participants will self-report how many times in the last 2 weeks they experienced symptoms from not at all to nearly every day.
Substance Use | Six Months
  We will assess participants alcohol and drug use via the SAMISS (Substance Use Subsection - AUDIT) questionnaire. Participants will self-report how many times a month they partake in alcohol or drug use on a scale ranging from never to less than monthly, to daily. Participants may also refuse to answer questions.
Wellness | Six Months
  We will assess participant's comprehensive health status measure using the Measure of Wellness (Medical Outcomes Study-HIV) survey. Participants will self-report how frequently they experienced symptoms relating to mental health, quality of life, health distress, cognitive function, energy/fatigue, overall health, role function, physical function, pain, and social function on a scale from all of the time to none of the time.
Stress | Six Months
  We will assess participant's ability to cope with stressful live events using the brief COPE self-report questionnaire. Participants will indicate how frequently they have utilized different coping mechanisms on a scale from not at all to a lot.
Resilience | Six Months
  We will assess participant's resilience using the Connor-Davidson Resilience Scale (CDRISC-100) self-report questionnaire. Participants will indicate the extent to which they identify with resilience statements from a scale from not at all true to true nearly all the time.
Implementation Factors | Six Months
  Acceptability, feasibility and appropriateness of our intervention will be quantitatively be measured as participants indicate how confident they feel in varying aspects of the intervention from not at all confident to completely confident.
Perceptions of Acceptability | Six Months
  Participant's views of the acceptability of our intervention will be measured using qualitative exit interviews.
Perceptions of Fidelity | Six Months
  The fidelity of our intervention will be measured using a fidelity monitoring tool. A research assistant (RA) will report yes, no, partially, or not applicable in response to statements about facilitators. The RA will also assess how well the facilitator did using a scale from poor to always.

CONTACTS AND LOCATIONS:
Locations (3):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- South Africa (2):
  - Desmond Tutu Health Foundation, East London, Eastern Cape
  - Desmond Tutu Health Foundation, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bondarchuk CP, Lemon T, Medina-Marino A, Rousseau E, Sindelo S, Sibanda N, Butler LM, Bekker LG, Earnshaw VA, Katz IT. A Moderated Mediation Model of HIV-Related Anticipated Stigma and Social Capital on the Relationship Between Diagnosis During the COVID-19 Pandemic and Potentially Problematic Substance Use Among Young South Africans. Int J Behav Med. 2025 Nov 18. doi: 10.1007/s12529-025-10415-5. Online ahead of print. PMID 41249762
- [Derived] Nardell MF, Sindelo S, Rousseau E, Siko N, Fuzile P, Julies R, Bassett IV, Mellins CA, Bekker LG, Butler LM, Katz IT. Development of "Yima Nkqo," a community-based, peer group intervention to support treatment initiation for young adults with HIV in South Africa. PLoS One. 2023 Jun 15;18(6):e0280895. doi: 10.1371/journal.pone.0280895. eCollection 2023. PMID 37319250